CLINICAL TRIAL: NCT05936515
Title: Evaluation of the Impact of a Paramedical Training Program for Nurses and Nursing Assistants on the Length of Stay and Prevention of Hospital Iatrogenic Complications in Elderly Patients
Acronym: CORRESPAGE
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 22-5125
Record Dates: First submitted 2023-06-22; First posted 2023-07-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-06

CONDITIONS: Iatrogenesis
Keywords: Care of the elderly; training of paramedical duo; specialtist wards; geriatric resource nurse
MeSH Terms: interventions — Nursing Assistants

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Post-intervention group (Training course group): The experimental group will be composed of patients aged 75 and over hospitalised in specialised departments after the establishment of geriatric correspondents trained in the specific care for the elderly.
  Interventions: Other: Training of nurses and nursing assistants
- Pre-intervention group (Control group): The control group will be composed of patients aged 75 years and over hospitalised in specialised departments before the introduction of geriatric correspondents trained in the specific care for the elderly. Their care will be conducted in accordance with usual practices.

INTERVENTIONS:
Other: Training of nurses and nursing assistants — Training of nurses and nursing assistants, based on the model of hygiene correspondents, in order to disseminate good geriatric practices
  Groups: Post-intervention group (Training course group)

SUMMARY:
In France, hospitalised elderly patients (EP) aged >75 years are expected to represent 1/3 of patients by 2030 (22% in 2015). In acute care wards outside geriatrics, the average length of stay increases with age, i.e. 8.5 days after the age of 90 compared with 5.5 days for younger patients. Dependence related to hospitalisation, partly avoidable, occurs in 30 to 60% of patients aged over 70. Faced with this situation Geriatric Mobile Teams (GMT) were created in 2002 to meet the need for geriatric expertise in hospitals and in the community by making punctual evaluations. Expert and multidisciplinary, the GMTs are a referring team for "advice, information and training for health care teams" for the care of vulnerable EPs. The GMTs are dependent on an exclusively medical demand system. The lack of knowledge of a specific care for EPs by nurses and nursing assistants and the occasional contribution of GMTs prevents a systematic targeted a for EP. Over the past 30 years, an American nursing programme (NICHE) aimed at improving the overall care of EPs in hospitals has shown that the training of geriatric resource nurses in speciality wards brought about a significant change in hospital geriatric culture. The training is based on evidence based practice including the HELP programme targeting confusion. The HELP programme has shown that nurses and nursing assistants play a pivotal role in reducing the incidence of hospital confusion. In the USA, the implementation of NICHE begins with the creation of a team of nursing leaders (geriatric/education/clinical care experts), dedicated to the coordination of the training and the companionship of geriatric resource nurses. Within the framework of the targets of the Ségur de la santé 2020 and Ma Santé 2022, our hypothesis is that an adaptation of NICHE to the French health context could improve specific care for EP in specialist wards, reduce the occurrence of complications and reduce the length of stay. Indeed, the GMT would ensure this coordination role in the training and support of a nurse and nursing assistant duo, based on the model of hygiene correspondents, in order to disseminate good geriatric practices.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 75 years and over hospitalised in a participating specialtist wards
* not objecting to the study,
* including those under guardianship or curatorship.

Exclusion Criteria:

* Patient not affiliated to a social security scheme
* Patient at the end of life

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: This study covers patients aged 75 and over hospitalised in participating specialitist wards (excluding geriatrics) (medicine, rheumatology, neurology, pneumology, orthopaedic surgery, digestive surgery, ENT and facial surgery)
Sampling Method: Non-Probability Sample
Enrollment: 2671 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Length of stay | The length of stay is calculated as the number of days between admission to the inclusion service and discharge documented in the medical record, assessed up to one month.
  Length of stay compared between groups according to whether or not geriatric correspondents are in place. This criterion has the advantage of being easy to measure, robust and a reflection of overall care. It depends on the occurrence of complications that can be prevented by the intervention of paramedical staff.

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Centre Hospitalier de Bourg en Bresse, Bourg-en-Bresse
  - Croix Rousse Hospital, Lyon
  - CH Annecy Genevois, Metz-Tessy
  - service de court séjour gériatrique, Hôpital Lyon Sud, Pierre-Bénite
  - Hôpital Nord-Ouest, Villefranche-sur-Saône